CLINICAL TRIAL: NCT03097614
Title: Prospective, Single-Arm Clinical Trial to Evaluate Acute Dry Eye Symptom Relief Assessed During Exposure to a Controlled Adverse Environment (CAE®) Following a 45 Day Period With Application of TrueTear™
Brief Title: Dry Eye Symptom Relief Assessment With Use of TrueTear in a Controlled Adverse Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oculeve, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCUN-029; NCT03180047 (obsolete NCT alias)
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Results first posted 2018-07-19 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-09

CONDITIONS: Dry Eye; Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TrueTear (Experimental): The device delivers small electrical currents, activating nerves that stimulate the body's natural tear production system.
  Interventions: Device: TrueTear

INTERVENTIONS:
Device: TrueTear — The device delivers small electrical currents, activating nerves that stimulate the body's natural tear production system.

SUMMARY:
This study characterizes acute dry eye symptom control, assessed during exposure to a Controlled Adverse Environment, following use of the TrueTear for 45 days.

DETAILED DESCRIPTION:
Subjects will be instructed to use the TrueTear daily for approximately 45 days with assessments in the Controlled Adverse Environment taking place on Day 0 and Day 45. Upon entering the CAE, participants will complete dry eye symptom questionnaires every five minutes and will administer the device when a certain level of ocular discomfort has been reached.

ELIGIBILITY:
Inclusion Criteria:

* Have used and/or desired to use an artificial tear substitute for dry eye symptoms within 6 months prior to the Screening Visit
* Normal lid/lash anatomy, blinking function and closure as determined by the Investigator
* Literate, able to speak English, and able to complete questionnaires independently

Exclusion Criteria:

* Chronic or recurrent epistaxis, coagulation disorders or other conditions that, in the opinion of the Investigator, may lead to risk of clinically significant increased bleeding
* Nasal or sinus surgery (including history of application of nasal cautery) or significant trauma to these areas
* Contact lens use within 7 days prior to the Screening Visit or anticipate the use of contact lenses at any time during the study
* Corneal transplant in either or both eyes
* Cardiac demand pacemaker, implanted defibrillator, or other active implanted metallic or active implanted electronic device in the head
* A woman who is pregnant, nursing an infant, or planning a pregnancy during the duration of the study
* Currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days prior to the Screening Visit

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, MD, Principal Investigator — Andover Eye Associates
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 57 enrolled subjects, 54 subjects completed the study. All 57 subjects enrolled in the study were included in FAS and safety populations
Period: Overall Study
Arm/Group | TrueTear
Started | 57
Completed | 54
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | TrueTear
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.3 (9.6)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 43
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 57
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Eye Dryness Score
Description: Eye Dryness Score using a visual analog scale assessed in the Controlled Adverse Environment (CAE). The participant rates their current eye dryness (both eyes simultaneously) by scoring 0 to indicate "no discomfort" and 100 to indicate "maximal discomfort". The assessment line length of the scale will be 100 mm.
Time Frame: Day 45
Population: Of the 57 subjects that initiated the study, 48 subjects achieved the threshold and performed an application in the CAE at Day 45.
Measure: Mean (Standard Error); unit: Score on Scale
Arm/Group | TrueTear
Number analyzed (Participants) | 48
Score on Scale | 48 (15.2)
Statistical Analysis 1: Comparison: TrueTear; Test type: Superiority; p = 0.0001, ANCOVA

ADVERSE EVENTS:
Time Frame: Day 45
Arm/Group | TrueTear
All-Cause Mortality (participants affected / at risk) | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57
Other Adverse Events (participants affected / at risk) | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study is the property of Allergan. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Allergan

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT03097614/Prot_SAP_000.pdf